CLINICAL TRIAL: NCT06753396
Title: Evaluation of the Effect of Injectable Platelet-Rich Fibrin on Peri-Implant Soft Tissue Phenotype
Brief Title: The Effect of Injectable Platelet-Rich Fibrin in Peri-implant Soft Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Berceste Guler, Associate Professor Dr., Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-17/08
Record Dates: First submitted 2024-11-26; First posted 2024-12-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Peri-Implant Tissues
Keywords: Peri-implant soft tissue; Injectable platelet-rich fibrin; Platelet-rich fibrin; Phenotype

STUDY DESIGN:
Intervention Model Description: The study will include 80 systemically healthy and non-smoking patients/implants older than 18 years of age with insufficient peri-implant keratinized mucosa width and mucosal thickness who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology. There are two study groups according to peri-implant mucosa phenotype: Thin phenotype and thick phenotype.-Thin phenotype: Mucosa thickness is less than 1 mm and the visibility of the probe in the sulcus is high.
  -Thick phenotype: Mucosa thickness is greater than 1 mm and visibility of the probe in the sulcus is low.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thin phenotype (Other): Mucosa thickness is less than 1 mm and the visibility of the probe in the sulcus is high.
  Interventions: Procedure: Platelet rich fibrin
- Thick phenotype (Other): Mucosa thickness is greater than 1 mm and visibility of the probe in the sulcus is low.
  Interventions: Procedure: Platelet rich fibrin

INTERVENTIONS:
Procedure: Platelet rich fibrin — The injectable platelet rich fibrin will be integrated into the tissue by subgingival and submucosal application to the keratinized gingiva of the implant sites with insufficient peri-implant soft tissue phenotype. Then, the prepared injectable platelet rich fibrin will be injected into the mucogingival junction apical to the keratinized gingival site. This procedure will be repeated 3 times in total, 1 time in 30 days for 3 months.
  Other Names: Injectable plateler rich fibrin

SUMMARY:
An inadequate amount of peri-implant soft tissue results in more plaque accumulation around the implants, peri-implant mucositis, marginal bone loss, mucosal recession, and/or attachment loss. In the literature, there are studies evaluating the application of injectable platelet-rich fibrin to the gingiva and oral mucosa around teeth, but injectable platelet-rich fibrin application around implants has not been encountered. This study aimed to evaluate the effect of subgingival and submucosal application of injectable platelet-rich fibrin on peri-implant soft tissue phenotype in patients with inadequate peri-implant soft tissue phenotype.The study will include 80 systemically healthy and non-smoking patients/implants older than 18 years of age with insufficient peri-implant keratinized mucosa width and mucosal thickness who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology. There are two study groups according to peri-implant mucosa phenotype: Thin phenotype and thick phenotype. All patients will undergo the same procedure of injectable platelet-rich fibrin application

DETAILED DESCRIPTION:
The peri-implant soft tissue phenotype comprises keratinized mucosal width mucosal thickness, and supracrestal tissue height. Peri-implant soft tissue has been at the center of debate for the last decade, playing a critical role in implant esthetics and peri-implant health. Various methods such as bone grafts, autologous soft tissue grafts, non-cellular dermal matrix, autologous platelet concentrates, and hyaluronic acid are used to increase the peri-implant soft tissue phenotype. Most of these methods are surgical and invasive. Recently, the use of autologous platelet concentrates has been proposed to support oral soft and hard tissue regeneration in regenerative periodontology and implant dentistry. Injectable platelet-rich fibrin from autologous platelet concentrates is a bioactive agent obtained by centrifugation at low speed. Its high content of white blood cells and high concentration of growth factors provide an important advantage for the regeneration process. It has been demonstrated that platelets release extracellular vesicles, which are thought to be necessary for tissue regeneration and can change the phenotype and function of recipient cells by carrying various proteins, bioactive lipids, and even genetic information through extracellular vesicles. In a study of 33 patients with thin gingival phenotype, injectable platelet-rich fibrin was applied on one side and injectable platelet-rich fibrin with microneedling on the other side, and mucosal thickness and keratinized mucosal width were compared. According to the results of the study, it was observed that mucosal thickness increased more in the group in which injectable platelet-rich fibrin was applied with the microneedling method. It was stated that microneedle application of injectable platelet-rich fibrin was less invasive and injectable platelet-rich fibrin showed good results in increasing mucosal thickness. In the literature, there are studies evaluating the application of injectable platelet-rich fibrin to the gingiva and oral mucosa around the tooth, but injectable platelet-rich fibrin application around the implant has not been encountered. To evaluate the effect of subgingival and submucosal injectable platelet-rich fibrin application on peri-implant soft tissue phenotype in patients with insufficient peri-implant soft tissue phenotype.

The study will include 80 systemically healthy and non-smoking patients/implants older than 18 years of age with insufficient peri-implant keratinized mucosal width and mucosal thickness who applied to Kütahya University of Health Sciences, Faculty of Dentistry, Department of Periodontology. Systemic and dental anamnesis will be taken from the patients before the operation, clinical measurements (plaque index, gingival index, clinical attachment loss, bleeding index on probing, pocket depth, peri-implant keratinized mucosa width, peri-implant mucosa thickness, and peri-implant gingival phenotype) will be recorded, standardized photographs will be obtained from the region and pink esthetic scoring will be performed. Implants with insufficient peri-implant soft tissue phenotype will be locally anesthetized. There are two study groups according to peri-implant mucosa phenotype: Thin phenotype and thick phenotype. Before the procedure, venous blood taken from the patient will be centrifuged at 700 RPM for 3 minutes in glass tubes without addition to obtain injectable platelet-rich fibrin. Injectable platelet-rich fibrin will be taken into a 2 cc syringe. The injectable platelet-rich fibrin will be integrated into the tissue by subgingival and submucosal application to the keratinized gingiva of the implant sites with insufficient peri-implant soft tissue phenotype. Then, the prepared injectable platelet-rich fibrin will be injected into the mucogingival junction apical to the keratinized gingival site. This procedure will be repeated 3 times in total, 1 time in 30 days for 3 months. Postoperatively, standardized photographs will be obtained at 1, 3, 6, and 12 months, pink esthetic scoring will be performed, and keratinized gingival height, keratinized mucosa width, mucosal thickness, and gingival phenotype will be recorded in the peri-implant site.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. The patient does not have any systemic disease
3. Patients who do not smoke or who smoke less than 10 cigarettes
4. Peri-implant keratinized mucosa width less than 2 mm
5. Peri-implant mucosal thickness less than 2 mm

Exclusion Criteria:

1. Being out of the defined age group
2. Any systematic contraindication for periodontal surgery
3. Patients who smoke more than 10 cigarettes per day
4. Patients with adequate peri-implant keratinized mucosa width and mucosal thickness
5. Pregnancy
6. Patients taking medication that suppresses the immune system or impairs healing
7. Patients taking medication that impairs the bleeding condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Peri-implant keratinized mucosa width | 1-year follow-up of all implants
  To measure peri-implant keratinized mucosa width of subgingival and submucosal injection of injectable platelet-rich fibrin in patients with inadequate peri-implant soft tissue phenotype at 1-year follow-up.
Peri-implant mucosa thickness | 1-year follow-up of all implants
  To measure peri-implant mucosa thickness of subgingival and submucosal injection of injectable platelet-rich fibrin in patients with inadequate peri-implant soft tissue phenotype at 1-year follow-up.

SECONDARY OUTCOMES:
Pink esthetic score | 1-year follow-up of all implants
  To measure the effect of subgingival and submucosal injectable platelet-rich fibrin application on the pink aesthetic score by the patient and physician in patients with inadequate peri-implant soft tissue phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler Ayyıldız, Assoc. Prof. Dr, Study Director — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP
Time Frame: The work will be shared 6 months after publication
Access Criteria: It will be shared in case the principal investigator is contacted.

REFERENCES:
- [Background] Faour NH, Dayoub S, Hajeer MY. Evaluation of the Hyaluronic Acid Versus the Injectable Platelet-Rich Fibrin in the Management of the Thin Gingival Phenotype: A Split-Mouth Randomized Controlled Clinical Trial. Cureus. 2022 May 18;14(5):e25104. doi: 10.7759/cureus.25104. eCollection 2022 May. PMID 35607316
- [Background] Ozsagir ZB, Saglam E, Sen Yilmaz B, Choukroun J, Tunali M. Injectable platelet-rich fibrin and microneedling for gingival augmentation in thin periodontal phenotype: A randomized controlled clinical trial. J Clin Periodontol. 2020 Apr;47(4):489-499. doi: 10.1111/jcpe.13247. Epub 2020 Feb 11. PMID 31912532
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Background] Frizzera F, Oliveira GJPL, Shibli JA, Moraes KC, Marcantonio EB, Marcantonio Junior E. Treatment of peri-implant soft tissue defects: a narrative review. Braz Oral Res. 2019 Sep 30;33(suppl 1):e073. doi: 10.1590/1807-3107bor-2019.vol33.0073. eCollection 2019. PMID 31576957
- [Background] Bouri A Jr, Bissada N, Al-Zahrani MS, Faddoul F, Nouneh I. Width of keratinized gingiva and the health status of the supporting tissues around dental implants. Int J Oral Maxillofac Implants. 2008 Mar-Apr;23(2):323-6. PMID 18548930
- [Background] Schrott AR, Jimenez M, Hwang JW, Fiorellini J, Weber HP. Five-year evaluation of the influence of keratinized mucosa on peri-implant soft-tissue health and stability around implants supporting full-arch mandibular fixed prostheses. Clin Oral Implants Res. 2009 Oct;20(10):1170-7. doi: 10.1111/j.1600-0501.2009.01795.x. Epub 2009 Aug 30. PMID 19719741
- [Background] Chung DM, Oh TJ, Shotwell JL, Misch CE, Wang HL. Significance of keratinized mucosa in maintenance of dental implants with different surfaces. J Periodontol. 2006 Aug;77(8):1410-20. doi: 10.1902/jop.2006.050393. PMID 16881810
- [Background] Tavelli L, Barootchi S, Avila-Ortiz G, Urban IA, Giannobile WV, Wang HL. Peri-implant soft tissue phenotype modification and its impact on peri-implant health: A systematic review and network meta-analysis. J Periodontol. 2021 Jan;92(1):21-44. doi: 10.1002/JPER.19-0716. Epub 2020 Aug 9. PMID 32710810